CLINICAL TRIAL: NCT04010916
Title: The Efficacy of Ultrasound-Guided Adductor Canal Block Timing for Postoperative Analgesia Management After Arthroscopic Knee Surgery
Brief Title: The Efficacy Of Ultrasound-Guided Adductor Canal Block for Arthroscopic Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol MH
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Knee Arthropathy
Keywords: Postoperative analgesia; Adductor canal block; Knee arthroscopy

STUDY DESIGN:
Intervention Model Description: Ninety patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for arthroscopic knee surgery will be included in the study. Patients will be randomly divided into three groups (Group Pre = preoperatively before inflation of the tourniquet group, Group Pre-T = preoperatively after inflation of the tourniquet group, Group Post = Postoperatively group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Pre = preoperatively before inflation of the tourniquet (Active Comparator): ACB will be performed under general anesthesia in the supine position. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit
  Interventions: Other: Group Preoperatively Adductor Canal Block
- Group Pre-T = preoperatively after inflation of the tourniquet (Active Comparator): ACB will be performed under general anesthesia in the supine position. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit
  Interventions: Other: Group Preoperatively Tourniquet Adductor Canal Block
- Group Post = Postoperatively group (Active Comparator): ACB will be performed under general anesthesia in the supine position. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit
  Interventions: Other: Group Postoperatively Adductor Canal Block

INTERVENTIONS:
Other: Group Preoperatively Adductor Canal Block — The ACB will be performed preoperatively before inflation of the tourniquet. After identifing the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be remowed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 30 mL will be injected here.
  Arms: Group Pre = preoperatively before inflation of the tourniquet
Other: Group Preoperatively Tourniquet Adductor Canal Block — The ACB will be performed preoperatively after inflation of the tourniquet. After identifing the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be remowed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 30 mL will be injected here.
  Arms: Group Pre-T = preoperatively after inflation of the tourniquet
Other: Group Postoperatively Adductor Canal Block — The ACB will be performed postoperatively. After identifing the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be remowed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 30 mL will be injected here.
  Arms: Group Post = Postoperatively group

SUMMARY:
The ultrasound-guided selective blockade of the saphenous nerve in the adductor canal provides effective analgesia and reduces postoperative pain in patients undergoing arthroscopic medial meniscectomy. Selective blockade of the saphenous nerve in the adductor canal provides effective analgesia without quadriceps muscle weakness. It has been shown that usage of tourniquet during performing the adductor canal block (ACB) block increases the spread of local anesthetics in a distal and proximal way. Therefore, the proximal spread of local anesthetics may cause possible quadriceps weakness. The distal spread of local anesthetics may increase analgesic effect via sciatic nerve. The timing of the tourniquet inflation for ACB is a topic of discussion.The aim of this study is to compare the different times of US-guided ACB performing for postoperative analgesia management after arthroscopic knee surgery.

DETAILED DESCRIPTION:
Knee arthroscopy is one of the most common orthopedic procedures. Knee arthroscopy is commonly used for the repairement of meniscus tears, debridement and reshaping of cartilage flaps, and ligament reconstruction. Knee arthroscopy is a minimally invasive procedure, however patients may complain severe pain due to the port-site incisions and the ligaments in the knee joint. Opioid agents are commonly used for analgesia management. However, opioids have adverse effects such as nausea, vomiting, sedation and respiratory depression. Peripheral nerve blocks such as femoral block, adductor canal block (ACB) may be performed to reduce opioid consumption and opioid-related side effects.

Selective blockadge of the saphenous nerve in the adductor canal for knee surgery provides effective analgesia without quadriceps muscle weakness. This is an important advantage of ACB since it there is no motor blockadge in the postoperative period. Blocking of the motor branches leads to delaying of the mobilization and it increases the patient's falling risk. ACB, targets the saphenous nerve and the vastus medialis branch which are the two largest sensorial nerves of the femoral nerve that innervates the knee. ACB blocks the articular branches of the obturator nerve at the same time. Since the ACB is performed at the distal site of thigh it does not target majority of the efferent branches of the quadriceps muscle, therefore the strength of this muscle may not be affected.

ACB is an effective and safely block. It has been shown that usage of the tourniquet during performing the ACB block increases the spread of local anesthetics in a distal and proximal way. There are two questions in this issue. Firstly, the proximal spread of local anesthetics may cause possible quadriceps weakness. Secondly the distal spread of local anesthetics may increase analgesic effect via sciatic nerve blockade. In the routine surgical procedure, at the beginning of the surgery a tourniquet is attached to the thigh and inflated following the induction of anesthesia. Then at the end of the procedure the tourniquet is deinflated and the patient is extubated. ACB may be performed preoperatively or postoperatively. It may be performed before or after the inflation of the tourniquet.

The aim of this study is to compare the different performing times of US-guided ACB for postoperative analgesia management after arthroscopic knee surgery. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), and adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for arthroscopic knee surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* Receiving anticoagulant treatment
* Known local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Postoperative 24 hours
  Fentanyl using

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative 24 hours period
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 0, 2, 4, 8, 16 and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Bahadir Ciftci, Asist.Prof, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Kejriwal R, Cooper J, Legg A, Stanley J, Rosenfeldt MP, Walsh SJ. Efficacy of the Adductor Canal Approach to Saphenous Nerve Block for Anterior Cruciate Ligament Reconstruction With Hamstring Autograft: A Randomized Controlled Trial. Orthop J Sports Med. 2018 Oct 10;6(10):2325967118800948. doi: 10.1177/2325967118800948. eCollection 2018 Oct. PMID 30345322
- [Background] Hanson NA, Derby RE, Auyong DB, Salinas FV, Delucca C, Nagy R, Yu Z, Slee AE. Ultrasound-guided adductor canal block for arthroscopic medial meniscectomy: a randomized, double-blind trial. Can J Anaesth. 2013 Sep;60(9):874-80. doi: 10.1007/s12630-013-9992-9. Epub 2013 Jul 3. PMID 23820968
- [Background] Jaeger P, Jenstrup MT, Lund J, Siersma V, Brondum V, Hilsted KL, Dahl JB. Optimal volume of local anaesthetic for adductor canal block: using the continual reassessment method to estimate ED95. Br J Anaesth. 2015 Dec;115(6):920-6. doi: 10.1093/bja/aev362. PMID 26582853